CLINICAL TRIAL: NCT02304757
Title: Prospective Trial of 99Tc-MDP and Fosamax in Postmenopausal Women With Differentiated Thyroid Cancer and Osteoporosis Treated With Supraphysiological Doses of Thyroid Hormone
Brief Title: 99Tc-MDP in Postmenopausal Women With Differentiated Thyroid Cancer and Osteoporosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Chao Ma, Dr., Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SanghaiXinhua
Record Dates: First submitted 2014-11-24; First posted 2014-12-02 (Estimated); Results first posted 2021-10-18 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Differentiated Thyroid Cancer; Osteoporosis
Keywords: differentiated thyroid cancer; bone mineral density; thyroid stimulating hormone suppression
MeSH Terms: conditions — Osteoporosis | interventions — Technetium; Alendronate

STUDY DESIGN:
Intervention Model Description: Patients with OS were divided into 99Tc-MDP and fosamax treatment groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 99Tc-MDP (Experimental): 15mg 99Tc-MDP were intravenously administered twice a week for 10 weeks, then once a week for 8 weeks, every two weeks for 22 weeks and monthly for another 3m.
  Interventions: Drug: 99Tc-MDP
- Fosamax (Active Comparator): 70mg po every week for 12 months.
  Interventions: Drug: Fosamax

INTERVENTIONS:
Drug: 99Tc-MDP — 99Tc-MDP, H20000218
  Other Names: Yunke,Technetium [99Tc] Methylenediphosphonate
  Arms: 99Tc-MDP
Drug: Fosamax — H20080172
  Other Names: alendronate sodium
  Arms: Fosamax

SUMMARY:
Postmenopausal women with differentiated thyroid cancer (DTC) taking suppressive doses of levothyroxine (L-T4) are thought to have accelerated bone loss and increased risk of osteoporosis. Therefore, the investigators try to investigate the effects of 99Tc-MDP,alendronate sodium in postmenopausal women with DTC under TSH suppression and osteoporosis.

DETAILED DESCRIPTION:
Differentiated thyroid cancer (DTC) has become one of the most common endocrine malignancies. According to American Thyroid Association (ATA) and Chinese Thyroid Association (CTA), most of DTC patients undergo total or near total thyroidectomy, radioiodine ablation and TSH (thyroid stimulating hormone) suppression. Osteoporosis (OS) and fractures are important comorbidities in patients with DTC, with potential negative impact on quality of life (QOL) and survival. The main determinant of skeletal fragility in DTC is the TSH suppression. Postmenopausal women with DTC under TSH suppression therapy are more vulnerable to OS. Technetium-99 methylene diphosphonate (99Tc-MDP) is a decay product of 99mTc-MDP (used for bone scintigraphy) and a novel bisphosphonates, which has been used in China for diseases like rheumatoid arthritis (RA), ankylosing spondylitis (AS) and osteochondral lesions of the talus, etc. However, as a member of bisphosphates, little attention has been paid to its anti-OS effect for DTC under TSH suppression.

ELIGIBILITY:
Inclusion Criteria:

(1) They were pathologically diagnosed with DTC including papillary or follicular carcinoma. (2) They received a near total thyroidectomy and radioiodine treatment. (3) TSH suppression should be at least one year before the study. (4) Bone mineral density (BMD) in lumbar spine and/or hip was tested by Dual-energy X-ray absorptiometry (DXA) at baseline, 6 month (m) and/or 12m follow up. 5) The diagnosis of osteoporosis was T-score ≤-2.5 SD at the lumbar spine, or hip.

Exclusion Criteria:

1. patients having medications for osteoporosis before TSH suppression treatment;
2. secondary osteoporosis ;
3. severe liver or kidney disease;
4. myelosuppression;
5. digestive disease;
6. long term use of immunosuppressive agent, estrogen or estrogen receptor modulators. This study was approved by the Institutional Review Board of Hospital Research Ethics. All the patients were fully acquainted with their treatment and consented to participate in the clinical trial.

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chao Ma, MD, Principal Investigator — Shanghai 10th People's Hospital
Locations (1):
- Nuclear Medicine Xinhua Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled in three centers (Tenth People's Hospital of Tongji University, Shanghai No. 4 People's Hospital and Xinhua Hospital School of Medicine Shanghai Jiaotong University) from January 2015 to December 2019.
Pre-assignment Details: In the total of 142 included patients, 70 were treated with 99Tc-MDP and 72 were treated with Fosamax.
Groups:
- Fosamax: 70mg po every week for 12 months.
  Alendronate Sodium: H20080172
Period: Overall Study
Arm/Group | 99Tc-MDP | Fosamax
Started | 70 | 72
Completed | 70 | 72
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 99Tc-MDP | Fosamax | Total
Number analyzed (Participants) | 70 | 72 | 142
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.29 (7.96) | 62.73 (7.24) | 63 (7)
Sex/Gender, Customized [Number; unit: participants]
  Sex: Female | 70 | 72 | 142
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  China | 70 | 72 | 142
TNM staging [Number; unit: number of participants] — T1N0-1, indicated participants had tumor ≤2 cm in greatest dimension, and with (N1) or without (N0)metastasis to lymph node; T2N0-1, tumor size >2 cm but ≤4 cm in greatest dimension, and with or without metastasis to lymph node; T3N0-1, tumor size >4 cm, and with or without metastasis to lymph node; TxNX, indicated participants had unknown tumor size and unknown metastasis to lymph node; TxN0-1, indicated participants had unknown tumor size, and with or without metastasis to lymph node; T1-2Nx, tumor ≤2 cm(T1) or >2 cm but ≤4 cm (T2), and unknown metastasis to lymph node.
  number of participants
    T1N0-1 | 35 | 39 | 74
    T2N0-1 | 6 | 5 | 11
    T3N0-1 | 4 | 9 | 13
    T4N0-1 | 18 | 12 | 30
    TxNx | 1 | 1 | 2
    TxN0-1 | 5 | 4 | 9
    T1-2Nx | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percent Change of Bone Mineral Density in Lumbar and Hip
Description: Percent change of bone mineral density in lumbar and hip by dual energy x-ray absorptiometry
Time Frame: baseline, 6 months, and 12 months
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | 99Tc-MDP | Fosamax
Number analyzed (Participants) | 70 | 72
percentage change
  Percentage change of lumbar spine at month 6 | 3.0 (6.6) | 3.2 (7.1)
  Percentage change of lumbar spine month 12 | 3.8 (10.9) | 5.1 (6.1)
  Percentage change of total hip at month 6 | 0.9 (7.7) | 4.9 (7.7)
  Percentage change of total hip at month 12 | 5.1 (17) | 4.6 (9.6)

2. Secondary Outcome: Bone Turnover Markers
Description: bone turnover markers including C-telopeptides of type I collagen (CTX), Type I N-procollagen terminal propeptide(PINP)
Time Frame: baseline and 12 months
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | 99Tc-MDP | Fosamax
Number analyzed (Participants) | 70 | 72
ng/ml
  PINP before treatment | 43.7725 (14.74802) | 29.255 (29.46603)
  PINP at 12months | 52.6422 (20.56123) | 20.56123 (25.34437)
  CTX before treatment | 0.4657 (0.25277) | 0.1526 (0.14138)
  CTX at 12months | 0.3707 (0.21062) | 0.1771 (0.16019)

3. Secondary Outcome: Health Related Quality of Life by 36-item Short Form Health Status Survey Questionnaire (0-100)
Description: The health related quality of life was measured by 36-item Short Form Health Status Survey questionnaire (SF-36). The minimum and maximum values were 0 and 100, respectively. Higher scores mean a better a better outcome.
  The questionnaire includes 36 items that can be classified into the following eight health status subscales: Physical Functioning, Physical Role Limitations, Bodily Pain, General Health Perception, Vitality, Social Functioning, Emotional Role Limitations, and Mental Health. A standardized Physical Component Summary and a standardized mental component score were calculated. The physical component summary and mental component summary represent the deviation from the reference population in Sweden. Higher scores mean a better a better outcome.
Time Frame: baseline, 6 months, and 12 months
Measure: Mean (Full Range); unit: scores on a scale
Arm/Group | 99Tc-MDP | Fosamax
Number analyzed (Participants) | 70 | 72
scores on a scale
  Physical component summary at baseline by 36-item Short Form Health Status Survey questionnaire | 61.4 [17.5 to 92.5] | 64.4 [30.5 to 87.5]
  Physical component summary at 6months by 36-item Short Form Health Status Survey questionnaire | 67.587 [14 to 100] | 69.09 [25.5 to 94.25]
  Physical component summary at 12months by 36-item Short Form Health Status Survey questionnaire | 69 [30.25 to 94.25] | 68 [40 to 92.25]
  Mental component score at baseline by 36-item Short Form Health Status Survey questionnaire | 65.7 [19.38 to 100] | 65.7 [34.88 to 95.88]
  Mental component score at 6months by 36-item Short Form Health Status Survey questionnaire | 69.0359 [14 to 100] | 66.24 [39.38 to 95]
  Mental component score at 12months by 36-item Short Form Health Status Survey questionnaire (0-100) | 69.2645 [15 to 100] | 67.087 [37.75 to 92.25]

4. Secondary Outcome: Side Effects
Description: A transient rash and phlebitis, gastrointestinal reaction.
Time Frame: 6 months, and 12 months
Measure: Number; unit: side effects
Arm/Group | 99Tc-MDP | Fosamax
Number analyzed (Participants) | 70 | 72
side effects
  abdominal pain | 0 | 2
  dyspepsia | 0 | 4

ADVERSE EVENTS:
Time Frame: Adverse event data were collected at 1year.
Arm/Group | 99Tc-MDP | Fosamax
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/72
Serious Adverse Events (participants affected / at risk) | 0/70 | 0/72
Other Adverse Events (participants affected / at risk) | 0/70 | 6/72
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 99Tc-MDP (N=70) | Fosamax (N=72)
upper gastrointestinal (GI) adverse events (Gastrointestinal disorders) | 0 (0) | 6 (72) — In the 6/72 patients with GI adverse events treated with alendronate, 2 cases had abdominal pain, 4 had dyspepsia.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-16): https://cdn.clinicaltrials.gov/large-docs/57/NCT02304757/Prot_SAP_000.pdf